CLINICAL TRIAL: NCT02567968
Title: A Randomized, Double-Blinded, Placebo-Controlled Study to Determine if Caffeine Citrate Accelerates Emergence From Anesthesia
Brief Title: A Study to Determine if Caffeine Accelerates Emergence From Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: IRB15-0897; 1R01GM116119-01 (NIH)
Record Dates: First submitted 2015-09-30; First posted 2015-10-05 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Anesthesia
MeSH Terms: interventions — Caffeine; caffeine citrate; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Anesthetized volunteers will be allowed to wake after injection of either saline (placebo control) or caffeine (15 mg/ kg). The time to wake will be measured.
  Interventions: Drug: Placebo Control
- Caffeine (Active Comparator): Anesthetized volunteers will be allowed to wake after injection of either saline (placebo control) or caffeine (15 mg/ kg). The time to wake will be measured.
  Interventions: Drug: Caffeine

INTERVENTIONS:
Drug: Caffeine — Anesthetized volunteers will be allowed to wake after injection of caffeine (15 mg/ kg). The time to wake will be measured.
  Other Names: Caffeine citrate
  Arms: Caffeine
Drug: Placebo Control — Anesthetized volunteers will be allowed to wake after injection of saline (placebo control). The time to wake will be measured.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
At present clinicians have no way to reverse anesthesia. Patients wake when their bodies clear the anesthetic. Most people wake quickly, but some do not. All patients have memory and other cognitive problems after waking from anesthesia. In studies on animals, the investigators observed that caffeine caused rats and mice to wake much more rapidly from anesthesia. This was true for all the animals tested. The investigators would like to see if this holds true in humans. Will caffeine accelerate waking from anesthesia? Will it reverse the cognitive deficits associated with anesthesia, after waking?

The investigators carried out a modest trial with 8 test subjects. Each volunteer was anesthetized twice. Each volunteer was anesthetized one time and received an infusion of saline (placebo control), without the aid of any other drugs and the other time the volunteer received an infusion of a relatively low dose of caffeine. The order of saline versus caffeine was randomized and the study was done in a double blind manner. We observed that emergence from anesthesia was significantly accelerated by the caffeine infusion. No adverse events were observed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25-40.
2. Male.
3. Normal healthy subject without systematic diseases or conditions.
4. Metabolic Equivalents of Functional Capacity >= 5.
5. Low risk for Obstructive Sleep Apnea (OSA) based on the screening test (STOP-bang score established by American Society of Sleep Apnea): Yes to > 3 items- high risk of OSA
6. No History of Arrhythmia (Baseline EKG will be obtained during the history and physical session), seizure, liver and kidney diseases.
7. BMI < 30 kg/m2.
8. No history of prior difficulty with anesthesia.
9. No personal or family history of malignant hyperthermia.
10. No history of any mental illness.
11. No history of drugs or alcohol abuse (urine drug screens required).
12. Subjects capable of giving consent.
13. Living less than 30 miles away from University of Chicago.
14. No history of seizure disorders.
15. No history of head trauma.

Exclusion Criteria:

1. Age <25 or >40.
2. Female.
3. ASA physical status > 1 (normal healthy subject without systematic diseases or conditions)
4. Metabolic Equivalents of Functional Capacity (METs) < 5.
5. High risks for Obstructive Sleep Apnea (OSA) based on the screening test (STOP-bang score established by American Society of Sleep Apnea): Yes to > 3 items- high risk of OSA
6. History Arrhythmia (Baseline EKG will be obtained during the history and physical session), seizure, liver and kidney diseases
7. BMI>30 kg/m2.
8. Prior difficulty with anesthesia.
9. Personal or family history of malignant hyperthermia.
10. History of any mental illness.
11. History of drugs or alcohol abuse (urine drug screens required)
12. Subjects capable of giving consent
13. Living more than 30 miles away from University of Chicago.
14. History of seizure disorders.
15. History of head trauma.

Ages: 25 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-08; Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Fox, PhD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Caffeine, Then Placebo: Participants first received Caffeine. After a washout period of 2 weeks, they then received Placebo.
- Placebo, Then Caffeine: Participants first received Placebo, and after 2-week washout period, then received Caffeine
Period: First Intervention
Arm/Group | Caffeine, Then Placebo | Placebo, Then Caffeine
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: Washout (2 Weeks)
Arm/Group | Caffeine, Then Placebo | Placebo, Then Caffeine
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Caffeine, Then Placebo | Placebo, Then Caffeine
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to either receive Caffeine then Placebo or Placebo then Caffeine
Arm/Group | All Study Participants
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3
  Black | 3
  Asian | 2
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Waking Time - Re-establishment of the Gag Reflex.
Description: The goal of the study is to determine whether caffeine speeds emergence from anesthesia. The time between terminating delivery of anesthetic and the subject starting to gag was measured. Anesthesia suppresses the gag reflex. Immediately after anesthetizing the test subject, a laryngeal mask airway (LMA) device was inserted into the test subject airway. After anesthesia was terminated and emergence from anesthesia was taking place, the gag reflex was re-established, and the LMA produced a "gag response" in all test subjects. This objective and unequivocal measurement constituted the "emergence" time for each subject. The "emergence" time was defined as the time between terminating the anesthesia and the test subject starting to gag.
Time Frame: followed from the end of anesthesia to gag reflex, up to 2 hours
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Placebo: Placebo Control: Anesthetized volunteers will be allowed to wake after injection of saline (placebo control).
- Caffeine: Caffeine: Anesthetized volunteers will be allowed to wake after injection of caffeine (15 mg/ kg).
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 8 | 8
minutes | 16.45 (3.9) | 9.57 (5.1)
Statistical Analysis 1: Comparison: Placebo vs Caffeine; Test type: Superiority; p = 0.002, paired t-test

2. Secondary Outcome: Cognitive Test1 - Visual Analog Scale --- Feel Good
Description: Normally patients receiving anesthesia exhibit significant cognitive problems for hours after anesthesia is terminated. The goal is to determine whether caffeine helps ameliorate the cognitive issues. Fifteen minutes after terminating anesthesia each subject was asked to complete a series of psychomotor tests, if they were able. Otherwise the testing started at 30 minutes. The tests were repeated every 15 minutes. The first test, a visual analog scale (VAS) test consisted of two 100-mm lines, each labelled with of "feel good" or "feel bad" displayed on a computer screen. Test subjects were asked to rate how they currently felt by placing a cursor on each of the line (0=not at all, 100=extremely). The test repeated every 15 minutes.
Time Frame: Test was given at 15, 30, 45, 60, 75, 90, 105 and 120 minutes after terminating anesthesia.
Population: Some participants could not be tested at the early timepoints due to not being fully awake etc.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 8 | 8
units on a scale
  15 minutes post-anesthesia: number analyzed (Participants) | 1 | 5
  15 minutes post-anesthesia | 29 (0) | 54.8 (22.4)
  30 minutes post-anesthesia: number analyzed (Participants) | 7 | 7
  30 minutes post-anesthesia | 48.1 (29.5) | 50.3 (25.4)
  45 minutes post-anesthesia | 50.9 (29.0) | 58.1 (26.5)
  60 minutes post-anesthesia | 62.8 (26.5) | 55.1 (27.5)
  75 minutes post-anesthesia | 60.0 (28.2) | 59.3 (25.9)
  90 minutes post-anesthesia | 61.5 (26.7) | 59.5 (25.7)
  105 minutes post-anesthesia | 66.3 (24.1) | 61.9 (24.3)
  120 minutes post-anesthesia | 66.0 (25.1) | 66.8 (27.7)

3. Secondary Outcome: Cognitive Test1 - Visual Analog Scale --- Feel Bad
Description: as for outcome 2
Time Frame: Test was given at 15, 30, 45, 60, 75, 90, 105 and 120 minutes after terminating anesthesia.
Population: Some participants could not be tested at the early timepoints due to not being fully awake etc.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 8 | 8
units on a scale
  15 minutes post-anesthesia: number analyzed (Participants) | 1 | 5
  15 minutes post-anesthesia | 6.0 (0) | 27.4 (24.2)
  30 minutes post-anesthesia: number analyzed (Participants) | 7 | 7
  30 minutes post-anesthesia | 17.9 (20.9) | 11.6 (13.3)
  45 minutes post-anesthesia | 13.0 (14.1) | 11.8 (14.7)
  60 minutes post-anesthesia | 9.8 (10.3) | 10.0 (12.2)
  75 minutes post-anesthesia | 6.0 (8.1) | 8.5 (12.0)
  90 minutes post-anesthesia | 7.0 (7.2) | 6.4 (7.4)
  105 minutes post-anesthesia | 6.6 (11.0) | 3.9 (4.3)
  120 minutes post-anesthesia | 4.3 (4.3) | 4.3 (6.5)

4. Secondary Outcome: Cognitive Test2 - Sternberg Test of Memory
Description: Normally patients receiving anesthesia exhibit significant cognitive problems for hours after anesthesia is terminated. The goal is to determine whether caffeine helps ameliorate the cognitive issues. The test was first applied at 15 minutes following anesthesia, if the subject was awake and then repeated every 15 minutes. In the Sternberg Test of Memory (STM) participants were asked to memorize a string of numbers. Afterwards, a computer would flash a series of random numbers on the screen and the participant was asked whether the number on the computer screen was part of the earlier string or not. In three rounds, participants were given a string of 2, then 4, then 6 numbers. The latency until the subject answered the question was monitored and this is the data summarized here.
Time Frame: Test was given at 15, 30, 45, 60 minutes after terminating anesthesia.
Population: Some participants could not be tested at the early timepoints due to not being fully awake etc.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 8 | 8
ms
  15 minutes post-anesthesia: number analyzed (Participants) | 1 | 5
  15 minutes post-anesthesia | 847 (0) | 1001.4 (182.8)
  30 minutes post-anesthesia: number analyzed (Participants) | 7 | 7
  30 minutes post-anesthesia | 908.9 (146.9) | 853.7 (176.0)
  45 minutes post-anesthesia | 791.1 (99.6) | 780.8 (127.7)
  60 minutes post-anesthesia | 734.4 (100.1) | 733.5 (84.1)

5. Secondary Outcome: Cognitive Test3 - Divided Attention Task
Description: Normally patients receiving anesthesia exhibit significant cognitive problems for hours after anesthesia is terminated. The goal is to determine whether caffeine helps ameliorate the cognitive issues. The test was first applied at 15 minutes following anesthesia, if the subject was awake and then repeated every 15 minutes. In the Divided Attention Task (DAT), participants were asked to fly an airplane over the center of a winding road with a joystick and simultaneously press a button whenever targets randomly flashed on the screen. The computer program tracked the root mean squared (RMS) deviation of the plane from the center of the road and the latency for pressing the trigger when the target appeared.
Time Frame: Test was given at 15, 30, 45, 60 minutes after terminating anesthesia.
Population: Some participants could not be tested at the early timepoints due to not being fully awake etc.
Measure: Mean (Standard Deviation); unit: mm away from optimal
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 8 | 8
mm away from optimal
  15 minutes post-anesthesia: number analyzed (Participants) | 1 | 5
  15 minutes post-anesthesia | 26.3 (0) | 38.2 (4.3)
  30 minutes post-anesthesia: number analyzed (Participants) | 7 | 7
  30 minutes post-anesthesia | 38.2 (19.9) | 29.8 (14.0)
  45 minutes post-anesthesia | 35.2 (25.3) | 29.1 (13.3)
  60 minutes post-anesthesia | 24.5 (9.5) | 23.4 (6.4)

6. Secondary Outcome: Bispectral Index
Description: A bispectral index (BIS) measurement system was employed to measure depth of anesthesia. Using electrodes attached to the forehead to measure EEG, BIS outputs a dimensionless number between 0 and 100 that is proportional to the brain concentration of anesthetic and is thereby proportional to an individual's level of consciousness (Greenwald S, Chiang HH, Devlin P, Smith C, Sigl J, Chamoun N: The Bispectral Index (Bis2.0) as a Hypnosis Measure. Anesthesiology 1994; 81: A477-a477). When the test subjects arrive, prior to anesthesia, their BIS values are in the range of 95 - 99. That corresponds to an awake and alert state. During anesthesia, most subjects are in the range of 20 - 40, corresponding to an anesthetized state. As the anesthetic wears off, the BIS values rise until they are back in the 95 - 99 range that they were prior to anesthesia. In particular, we wished to determine whether BIS exhibited more rapid recovery after caffeine infusion as compared to saline (control).
Time Frame: Continuous monitoring from start of anesthesia until discharge of test subject, up to 2 hours post-anesthesia.
Population: One subject was missing data at the last timepoint for the Placebo session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 8 | 8
units on a scale
  0 minutes post-anesthesia | 34.1 (3.8) | 36.3 (3.5)
  2 min post-anesthesia | 41.4 (5.6) | 43.1 (15.4)
  4 min post-anesthesia | 48.5 (11.9) | 55.5 (13.8)
  6 minutes post-anesthesia | 55.0 (10.6) | 58.1 (11.7)
  8 minutes post-anesthesia | 60.3 (7.9) | 69.1 (11.7)
  10 minutes post-anesthesia | 62.5 (8.0) | 71.3 (9.5)
  12 minutes post-anesthesia | 62.9 (11.5) | 76.5 (12.5)
  14 minutes post-anesthesia | 62.6 (10.7) | 82.4 (11.2)
  16 minutes post-anesthesia: number analyzed (Participants) | 7 | 8
  16 minutes post-anesthesia | 69.1 (14.2) | 84.1 (11.9)

7. Secondary Outcome: Minute Ventilation
Description: The volume of gas inhaled or exhaled from a person's lungs per minute. We wished to determine whether caffeine altered minute ventilation.
Time Frame: Continuous monitoring from time lma inserted until subject started to gag and it was removed, up to 2 hours post-anesthesia.
Measure: Mean (Standard Deviation); unit: L/minute
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 8 | 8
L/minute
  Post-infusion | 6.2 (1.4) | 7.2 (1.1)
  Emergence | 7.5 (2.1) | 8.5 (3.7)

8. Secondary Outcome: Mean Arterial Blood Pressure
Description: This measurement was made in order to determine whether caffeine altered blood pressure in a deleterious manner.
Time Frame: Continuous monitoring from start of anesthesia until discharge of test subject, up to 2 hours post-anesthesia.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 8 | 8
mmHg
  Pre-anesthesia | 89 (9) | 90 (7)
  5 minutes after anesthesia | 72 (9) | 79 (15)
  30 minutes after anesthesia | 94 (10) | 98 (8)
  60 minutes after anesthesia | 96 (6) | 98 (6)

9. Secondary Outcome: Heart Rate
Description: This measurement was made in order to determine whether caffeine altered heart rate in a deleterious manner.
Time Frame: Continuous monitoring from start of anesthesia until discharge of test subject, up to 2 hours post-anesthesia.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 8 | 8
beats per minute
  Pre-anesthesia | 79 (13) | 75 (11)
  5 minutes after anesthesia | 71 (16) | 66 (10)
  30 minutes after anesthesia | 79 (7) | 75 (9)
  60 minutes after anesthesia | 67 (6) | 67 (9)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Placebo | Caffeine
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT02567968/Prot_SAP_001.pdf